CLINICAL TRIAL: NCT01383538
Title: A Phase I Study of FOLFIRINOX Plus IPI-926 for Advanced Pancreatic Adenocarcinoma
Brief Title: FOLFIRINOX Plus IPI-926 for Advanced Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew Ko (Other)
Collaborators: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Andrew Ko, Associate Professor, Department of Medicine (Hematology/Oncology), UCSF, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC#11455
Record Dates: First submitted 2011-06-20; First posted 2011-06-28 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cancer; Adenocarcinoma; Pancreatic Neoplasms
Keywords: pancreas; cancer; adenocarcinoma; Oxaliplatin; Leucovorin; Irinotecan; 5-FU; IPI-926
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Neoplasms | interventions — folfirinox; IPI-926; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRINOX Plus IPI-926 (Experimental)
  Interventions: Drug: FOLFIRINOX, IPI-926

INTERVENTIONS:
Drug: FOLFIRINOX, IPI-926 — Oxaliplatin: intravenous, 50 to 85 mg/m2, over 2 hrs, once per cycle.
  Leucovorin: intravenous, 400 mg/m2, over 2 hrs, once per cycle.
  Irinotecan: intravenous, 120 to 180 mg/m2, over 90 minutes, once per cycle.
  5-FU: intravenous, 1600 to 2400mg/m2, over 46hr continuous infusion, once per cycle.
  IPI-926: oral, 130 to 160 mg/day, daily, 14 days per cycle.
  Other Names: Oxaliplatin; Leucovorin; Irinotecan; 5-FU

SUMMARY:
The purpose of this phase I study to determine the optimal dose for the combination of IPI-926 plus FOLFIRINOX (5-fluorouracil, Leucovorin, Irinotecan, and Oxaliplatin) chemotherapy in patients with pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) represents the fourth leading cause of cancer-related mortality in the United States, with an estimated 36,800 deaths attributable to PDAC in 2010.(1) Over 90% of patients have inoperable disease at presentation, at which point systemic therapy becomes the primary form of treatment. Single agent gemcitabine became the standard of care for advanced pancreatic cancer a decade ago since demonstrating improved survival when compared with fluorouracil. Since then, a number of phase III trials have evaluated the benefit of adding additional cytotoxic or targeted agents to gemcitabine, as shown in the table below. The PA.3 trial(2), which led to the approval of erlotinib in advanced pancreatic cancer, was a landmark study in that it represented the first positive phase III study of a combination regimen for this disease indication; however, while erlotinib represents both an important proof of principle and a welcome addition to our therapeutic armamentarium, it has failed to gain significant traction in this disease, as many in the oncology community consider the marginal absolute improvement in median overall survival to be of questionable clinical significance.

FOLFIRINOX: A new standard of care for advanced PDAC? At the 2010 American Society of Clinical Oncology Annual Meeting (ASCO), a French cooperative group presented results of a potentially practice-changing phase III clinical trial (PRODIGE 4/ACCORD 11).(18) In this study, 342 patients with previously untreated metastatic pancreatic cancer were randomized to receive either gemcitabine monotherapy or the combination of biweekly infusional 5-fluorouracil, leucovorin, irinotecan, and oxaliplatin (FOLFIRINOX) (ref). The investigators reported statistically significant improvements for the FOLFIRINOX arm in the primary endpoint, overall survival (median of 11.1 months vs 6.8 months, P < .0001); as well as 1-year survival rate (48.4% vs. 20.6%), median progression-free survival (6.4 vs. 3.3 months; P < .0001), and objective response rate (CR+PR, 31.6% vs. 9.4%; P = .0001)). Not surprisingly, the more complex FOLFIRINOX regimen was associated with higher rates of grade 3/4 toxicities, including neutropenia (45.7% vs 18.7%), febrile neutropenia (5.4% vs. 0.6%), fatigue (23.2% vs. 14.2%), and diarrhea (12.7% vs. 1.2%). Notably, while primary prophylaxis with growth factor support was not mandated in this trial, 42.5% of patients did ultimately receive such support. Moreover, most patients enrolled in this trial had non-pancreatic head tumors (approximately 64%) which is the opposite distribution of what one might expect in a representative pancreatic cancer population. Thus, it is conceivable that the FOLFIRINOX regimen, with its high rates of neutropenia, may lead to unacceptable rates of infectious complications (eg, ascending cholangitis and biliary sepsis), in patients with pancreatic head tumors with indwelling endobiliary stents.

Nevertheless, this strikingly positive survival benefit, with a median overall survival approaching one year in a purely metastatic cohort, has never before been observed in any previous study, which raises the question of whether FOLFIRINOX should become the newly adopted standard of care, at least in patients with preserved performance status (patients on this trial were required to have an ECOG performance score of 0-1).

HEDGEHOG SIGNALING The Hedgehog(19) signaling pathway is important for normal mammalian embryonic development and for adult tissue remodeling. Recent reports have demonstrated that aberrant activation of the Hh pathway is associated with many types of cancer, including basal cell carcinoma (BCC), medulloblastoma, pancreatic adenocarcinomas, small-cell lung cancer (SCLC), metastatic prostate cancer, glioma, breast cancer, hepatocellular cancer, and hematologic malignancies. High levels of Hh pathway activation, either through mutation of pathway components or through constitutive expression of Hh pathway genes, appear to be involved in both the initiation of cancer and tumor cell survival, as well as tumor growth and metastasis. Given the therapeutic potential of Hh pathway inhibition in cancer, Infinity has developed IPI-926, a potent and specific antagonist of the Hh pathway that binds Smoothened (Smo), a key signaling transmembrane protein in this pathway, thereby diminishing downstream promoters of cellular proliferation.

Pancreatic adenocarcinomas are an ideal tumor class in which to evaluate the activity of a Hh pathway inhibitor, as multiple lines of evidence support a role for Hedgehog signaling in pancreatic tumorigenesis:

* Aberrant expression of Sonic hedgehog (SHH) and its associated signaling components (patched (PTC) and smoothened (SMO)) are frequently found in pancreatic cancer specimens.(20-27)
* Pharmacologic inhibition of hedgehog signaling produces antitumor effects in pancreatic cancer cell lines27 and orthotopic xenograft models.(28,29) Studies involving global sequencing analysis have identified this pathway as one of the central elements undergoing transformation in nearly all pancreatic cancers.(21)
* Hedgehog signaling may play an important role in maintenance of pancreatic cancer stem cells.(30-32)
* The dense desmoplastic mesenchymal network that constitutes the stroma of pancreatic adenocarcinomas coupled with poor vascularity may present a major challenge to effective delivery of intravenous chemotherapy to the bulk of pancreatic tumor cell burden. Recent evidence in a genetically engineered mouse model of pancreatic cancer demonstrated that IPI-926 can deplete tumor-associated stromal tissue and increase intratumoral mean vessel density, resulting in enhanced delivery of concurrently administered systemic agents such as gemcitabine, decreased tumor burden, and prolonged survival.(33)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed pancreatic adenocarcinoma
2. Disease that is not operable (locally advanced or metastatic)
3. No prior systemic therapy for their diagnosis (except in adjuvant setting > 6 months previously)
4. ECOG performance score of 0-1
5. At least 18 years of age
6. Evidence of either or both of the following:

   * RECIST-defined measurable disease (lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20mm using conventional techniques or ≥10 mm with spiral CT scan)
   * An elevated serum CA19-9 at baseline ( ≥ 2X ULN)
7. Endobiliary stents, but not percutaneous biliary drains, are permissible.
8. Adequate bone marrow function:

   * ANC ≥ 1500/uL
   * platelet count ≥ 100,000/uL
   * hemoglobin ≥ 9.0 g/dL (may be increased to this level with transfusion as long as there is no evidence of active bleeding)
9. Adequate hepatic function:

   * Total bilirubin ≤ 1.5 X ULN
   * AST (SGOT) ≤ 2.5 X ULN
   * ALT (SGPT) ≤ 2.5 X ULN
10. Adequate renal function as determined by either:

    * Calculated or measured creatinine clearance ≥ 40 mL/min (for calculated creatinine clearance, Cockcroft-Gault equation will be used). The Modified Cockcroft-Gault formula is as follows:

      [140 - age(yrs)] x [actual weight (kg)] / [72 x serum creatinine (mg/dl)] Note: Multiply by a factor of 0.85 if female
    * Serum creatinine ≤ 1.5 X ULN
11. Ability to swallow oral medications
12. All women of child-bearing potential (WCBP), all sexually active male patients, and all partners of patients must agree to use adequate methods of birth control throughout the study. Women of child-bearing potential (defined as being less than 1 year post-menopausal) must have a negative serum or urine β human chorionic gonadotropin (βhCG) pregnancy test; and men and women of reproductive potential must agree to practice an effective method of avoiding pregnancy while receiving study drug and for 30 days after the final dose of study drug. Effective contraception includes use of oral contraceptives with an additional barrier method, double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera, partner vasectomy, and total abstinence.
13. Ability to understand the nature of this study protocol and give written informed consent
14. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Any prior systemic or investigational therapy for metastatic pancreatic cancer. Systemic therapy administered alone or in combination with radiation in the adjuvant setting is permissible as long as it was completed > 6 months prior to the time of study enrollment.
2. Inability to comply with study and/or follow-up procedures.
3. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that, in the opinion of the investigator, renders the subject at high risk from treatment complications or might affect the interpretation of the results of the study.
4. Presence of central nervous system or brain metastases.
5. Life expectancy < 12 weeks
6. Pregnancy (positive pregnancy test) or lactation.
7. Concurrent active malignancy. The following prior malignancies ARE allowed: adequately treated non-melanoma skin cancer; in situ cervical cancer; localized prostate cancer; or adequately treated Stage I or II cancer for which treatment was completed more than one year ago and from which the patient is currently in complete remission; or any other form of cancer from which the patient has been disease-free for 5 years.
8. Patients with a history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months.
9. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
10. Known, existing uncontrolled coagulopathy. Patients who have had a venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation are eligible IF: they are appropriately anticoagulated and have not had a Grade 2 or greater bleeding episode in the 3 weeks before Day 1. However, as concurrent/pre-existing use of coumadin is not allowed, only low-molecular heparin should be used.
11. Pre-existing sensory neuropathy > grade 1.
12. Major surgery within 4 weeks of the start of study treatment, without complete recovery.
13. Cirrhotic liver disease, ongoing alcohol abuse, or known chronic active or acute hepatitis.
14. Concurrent administration of the medications or foods which are known to inhibit CYP3A activity to a clinically relevant degree (see Appendix 1).
15. Known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
16. Known hypersensitivity reaction to a sulfonamide.
17. Presence of active infection requiring systemic use of antibiotics within 72 hours of treatment.
18. Known human immunodeficiency virus (HIV) positivity.
19. Known hypersensitivity to IPI-926 or any of the excipients in IPI-926 capsules.
20. Pregnant or lactating women.
21. Any other co-morbid condition(s) that may interfere with study participation which in the judgment of the Investigator would place the patient at undue risk or interfere with the study. Examples include, but are not limited to sepsis, recent significant traumatic injury, and other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-08-23 (Actual); Primary Completion 2012-12-13 (Actual); Study Completion 2015-05-26 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) for FOLFIRINOX plus IPI-926 in patients with advanced pancreatic cancer. | Ongoing evaluation through sequential dose cohorts; evaluations at 2-week intervals up to one year.

SECONDARY OUTCOMES:
Number of participants with Adverse events and SAEs | Ongoing evaluation for all patients throughout the course of treatment; evaluations at 2-week intervals up to one year.
Time to tumor progression | Efficacy evaluations at 2-month intervals up to one year.
Objective response rate (ORR) by RECIST criteria | Efficacy evaluations at 2-month intervals up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, M.D., Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin